CLINICAL TRIAL: NCT05238077
Title: Comparing the Efficacy of VL-UVA1 Versus NB-UVB on Inducing Repigmentation in Subjects With Generalized Vitiligo
Brief Title: Comparing the Efficacy of Visible Light-Ultraviolet A1 Light Versus Narrowband-Ultraviolet B on Generalized Vitiligo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: only one subject enrolled, decided to re-evaluate protocol design
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Director Investigator Initiated Studies, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11973
Record Dates: First submitted 2019-07-22; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Generalized Vitiligo

STUDY DESIGN:
Intervention Model Description: The subject serves as their own control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VL-UVA1 vs NB-UVB (Other): Participants will be treated with both VL-UVA and NB-UVB on different areas
  Interventions: Procedure: Visible Light-Ultraviolet A Light or Narrowband-Ultraviolet B phototherapy

INTERVENTIONS:
Procedure: Visible Light-Ultraviolet A Light or Narrowband-Ultraviolet B phototherapy — Patients will have different kinds of light shined on different areas

SUMMARY:
As part of this study, you may have a procedure called phototherapy which involves either VL-UVA or NB-UVB irradiation. NB-UVB phototherapy is not experimental in vitiligo, but use of VL-UVA1 phototherapy in vitiligo is.

The purpose of this pilot study is to determine whether VL-UVA1 or NB-UVB phototherapy more efficiently induces repigmentation in patients with generalized vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age with a diagnosis of generalized vitiligo
* Subjects on a stable topical/oral regimen for the past 3 months and continuing on a stable regimen
* Subjects able to understand the requirements of the study
* Subjects able and willing to sign informed consent

Exclusion Criteria:

* Subjects on photosensitizing medications
* Subjects receiving any concurrent phototherapy
* Subjects who plan to use tanning parlors or expose themselves to excess sunlight
* Subjects with known photosensitivity disorder
* Subjects with apparent phototoxicity
* Subjects with unstable vitiligo
* Subjects currently using bleaching agents
* Subjects who are pregnant, lactating, or planning on becoming pregnant
* Subjects who in the opinion of the investigator/sub-investigator, are not appropriate candidates for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Change in depigmentation of vitiligo lesion | 13 measurements over 26 visits
  Change in pigment will be assessed by colorimetry which measures change in pigment
Change in melanin content of vitiligo lesion | 13 measurements over 26 visits
  Change in pigment will be assessed by diffuse reflectance spectroscopy which will measure the melanin content and dyschromia

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, M.D., Principal Investigator — Henry Ford HS
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No